CLINICAL TRIAL: NCT02886221
Title: Functional and Radiographic Outcomes of Hallux Valgus Correction by Mini-invasive Surgery With Reverdin-Isham Percutaneous Osteotomy: a Longitudinal Prospective Study With a 48-month Follow-up
Brief Title: Functional and Radiographic Outcomes of Hallux Valgus Correction by Mini-invasive Surgery With Reverdin-Isham Percutaneous Osteotomy
Acronym: MISHV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Carlo Biz, MD, Assistant Professor, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIS01
Record Dates: First submitted 2016-08-23; First posted 2016-09-01 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Hallux Valgus
Keywords: Hallux Valgus; Reverdin-Isham Osteotomy; Minimally Invasive Surgery; Percutaneous Distal Osteotomy; First Ray; Forefoot
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HV patients (Other): patients with symptomatic Hallux Valgus treated my Reverdin-Isham Osteotomy
  Interventions: Procedure: Reverdin-Isham Osteotomy

INTERVENTIONS:
Procedure: Reverdin-Isham Osteotomy — Incision on the medial part of the foot, a Shannon Isham burr was introduced at the junction of metaphysis and epiphysis. It was applied to the flat bone surface achieved previously at approximately 45°, keeping the articular cartilage surface of the first metatarsal head as reference point on the superior cortex. In this position, under fluoroscopic control, the osteotomy was started following a distal-dorsal and proximal-plantar direction. At this point, the burr was slightly withdrawn in order to preserve a few millimetres of the lateral cortex, and the osteotomy of the plantar cortex was performed completely. Then, a Wedge burr was used to create a wedge with a medially oriented base. At the point of closing the wedge, osteoclasis of the preserved lateral cortex was achieved, modifying the orientation of the articular surface, normalizing the DMAA value, and adding an intrinsic stability to the osteotomy by producing contact of the trabecular bone.

SUMMARY:
Minimally invasive surgery (MIS) represents one of the most innovative surgical treatments of Hallux Valgus (HV). However, long-term outcomes still remain a matter of discussion within the orthopaedic community. The purpose of this longitudinal prospective study was to evaluate radiographic and functional outcomes in patients with mild-to-severe HV who underwent Reverdin-Isham and Akin percutaneous osteotomy, following exostosectomy and lateral release.

DETAILED DESCRIPTION:
One hundred and eighty patients with mild-to-severe symptomatic HV were treated by MIS. Clinical evaluation was assessed pre-operatively, as well as at 3 and 12 months after surgery and at final follow-up of 48 months, using the American Orthopaedic Foot and Ankle Society (AOFAS) Hallux grading system. Patient satisfaction and complications were recorded.Further parameters assessed were postoperative pain at rest and during movement by the numerical rating scale (NRS), patient satisfaction using the Visual Analogue Scale (VAS), quality of life, and return to daily activities. Incidence of Chronic Pain Syndrome (CPS), Type of anesthesia and ASA were evaluated and recorded.

Computer-assisted measurement of antero-posterior radiographs was taken pre-operatively, as well as at 3 and 12 months after surgery and at 48-month follow-up, analysing the intermetatarsal angle (IMA), the hallux valgus angle (HVA), the distal metatarsal articular angle (DMAA), and the tibial sesamoid position. Also, the bridging bone/callus formation was evaluated at the different radiographic follow-ups, while the articular surface congruency and the metatarsal index were calculated only preoperatively and at last follow-up. Statistical analysis was carried out using the paired t-test. Statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to severe symptomatic hallux valgus

Exclusion criteria:

* congenital deformities of the foot
* hallux rigidus
* previous first ray trauma or foot and ankle surgery
* rheumatic, dismetabolic, neurologic, infective, or psychiatric pathologies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-05; Primary Completion 2020-06 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
clinical changes after surgical treatment | preoperative and at 3-12-48 months post-operative
  evaluation scale: AOFAS score

SECONDARY OUTCOMES:
radiological changes after surgical treatment | preoperative and at 3-12-48 months post-operative
  evaluation of the Intermetatarsal angle(IMA) of the first ray, distal metatarsal articular angle of the first metatarsal (DMAA), hallux valgus angle (HVA) and tibial sesamoid position
Postoperative pain levels and incidence of Chronic Pain Syndrome (CPS) | Patients were evaluated prospectively at 7 days, 1, 3 and 6 months after surgery for pain at rest and during movement.
  The parameters assessed were postoperative pain at rest and during movement by the numerical rating scale (NRS), patient satisfaction using the Visual Analogue Scale (VAS), quality of life, and return to daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Carlo Biz MD, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: Yes
Age, Gender, Radiological parameters and images.

REFERENCES:
- [Result] Mann RA, Coughlin MJ. Hallux valgus--etiology, anatomy, treatment and surgical considerations. Clin Orthop Relat Res. 1981 Jun;(157):31-41. PMID 7249460
- [Result] Trnka HJ. Osteotomies for hallux valgus correction. Foot Ankle Clin. 2005 Mar;10(1):15-33. doi: 10.1016/j.fcl.2004.10.002. PMID 15831256
- [Result] Isham SA. The Reverdin-Isham procedure for the correction of hallux abducto valgus. A distal metatarsal osteotomy procedure. Clin Podiatr Med Surg. 1991 Jan;8(1):81-94. PMID 2015537
- [Derived] Biz C, de Iudicibus G, Belluzzi E, Dalmau-Pastor M, Bragazzi NL, Funes M, Parise GM, Ruggieri P. Prevalence of chronic pain syndrome in patients who have undergone hallux valgus percutaneous surgery: a comparison of sciatic-femoral and ankle regional ultrasound-guided nerve blocks. BMC Musculoskelet Disord. 2021 Dec 15;22(1):1043. doi: 10.1186/s12891-021-04911-4. PMID 34911525
- [Derived] Biz C, Fosser M, Dalmau-Pastor M, Corradin M, Roda MG, Aldegheri R, Ruggieri P. Functional and radiographic outcomes of hallux valgus correction by mini-invasive surgery with Reverdin-Isham and Akin percutaneous osteotomies: a longitudinal prospective study with a 48-month follow-up. J Orthop Surg Res. 2016 Dec 5;11(1):157. doi: 10.1186/s13018-016-0491-x. PMID 27919259